CLINICAL TRIAL: NCT06071598
Title: The Role of Lipid Transporter MFSD2A in the Resolution of Colorectal Cancer-associated Inflammation: Implications for New Therapeutic Strategies
Brief Title: The Role of Lipid Transporter MFSD2A in the Resolution of Colorectal Cancer-associated Inflammation
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Silvio Danese, Director of Gastroenterology and Endoscopy Unit, IRCCS San Raffaele
Other Study IDs: CRCM 1.0
Record Dates: First submitted 2023-09-25; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CRC: CRC-affected patients stratified according to tumor stage (T0/T1-T4, M0/M1, N0/N1/N2)
  Interventions: Other: Surgical specimens of CRC-affected patients

INTERVENTIONS:
Other: Surgical specimens of CRC-affected patients — Specimens of CRC-affected patients will be collected during the surgery, without other risks for the patients, since we will use only material left after pathologist analysis

SUMMARY:
The intrinsic connection between inflammation and tumor promotion is well characterized and is a key pathogenic event in patients with colorectal cancer (CRC), the second most common cause of tumor-related death in western countries. Environmental factors and chronic inflammation represent the major causes of intestinal carcinogenesis. In fact, patients suffering from inflammatory bowel diseases, including Crohn's disease and Ulcerative Colitis (UC), have high risk of developing colitis-associated CRC with poor prognoses. Therefore, targeting the cancer-associated inflammation may offer new avenues for cancer treatment. In fact, several anti-inflammatory drugs, have been used for prophylaxis and have shown efficacy in contrasting cancer, despite various adverse side effects. Thus, there is an urgent need to discover novel cancer-associated mechanisms to develop alternative therapies that may reduce aberrant inflammatory responses without interfering with physiological defenses against infection and functional anti-tumor immunity. A novel approach promoting anti-tumor immunity has been recently proposed after the discovery of potent, endogenous, specialized pro-resolving mediators (SPMs), including lipoxins, resolvins, protectins, and maresins, mainly derived from omega-3 polyunsaturated fatty acid (PUFA) docosahexaenoic acid (DHA) and eicosapentaenoic acid (EPA) via COX, LOX and CYP450 pathways, mediated by MFSD2A. Due to the potent bioactivity of SPMs in resolving inflammation and because of the correlation between inflammation and cancer, the roles of these lipid mediators have attracted great attention for their potential therapeutic role in cancer treatment, including CRC. Nevertheless, the understanding of the endogenous mechanisms that limit the inflammatory response during CRC development is incomplete and requires further investigation.

Based on the preliminary results indicating that dysfunctional MFSD2A-dependent pro-resolving pathways may foster CRC development, the investigators aim to define the functional role of MFSD2A in orchestrating pro-resolving pathways in the intestinal endothelium of metastatic and not metastatic CRC patients.

This is a cross-sectional single-center observational study involving patients with CRC. The investigators will enroll 15 patients with colorectal cancer (CRC) stratified by tumor stage (T0 / T1-T4, M0 / M1, N0 / N1 / N2) undergoing surgery in the Gastroenterology and Digestive Endoscopy unit within Gastro Center (IRCCS Ospedale San Raffaele).

Human Intestinal Microvascular Endothelial Cells (HIMEC) will be generated from each sample of cancer surgical specimens, while the healthy cells will be derived from the healthy margins of the colorectal resection of the same CRC patients.

MFSD2A will be overexpressed or silenced and the investigators will evaluate its biological effects in both tumor-derived HIMECs and healthy tissue-derived HIMECs through transcriptomics and lipidomics analysis. The investigators will also exploit a possible novel therapy based on the delivery of MFSD2A encoding plasmid-conjugated liposomes.

ELIGIBILITY:
Inclusion Criteria:

- 15 CRC-affected patients stratified according to tumor stage (T0/T1-T4, M0/M1, N0/N1/N2)

Exclusion Criteria:

Patients:

* taking trace elements, hypolipemiants in the previous 3 months
* undergone previous intestinal resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To define the MFSD2A-dependent pro-resolving pathways and the relative production of lipid mediators in patients with metastatic CRC, CRC HIMEC will be isolated from surgical specimens of CRC-affected patients stratified according to tumor stage (T0/T1-T4, M0/M1, N0/N1/N2) (n=5/stage, CRC-HIMEC), while the healthy cells will be derived from the healthy margins of the colorectal resection of the same CRC patients.
  The participation is voluntary and the patient is allowed to refuse further participation in the protocol whenever he/she wants.
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
To define the functional role of MFSD2A in CRC through Polyunsaturated fatty acid (PUFA) ad genes analysis. | 1-36 months
  In particular, PUFAs will be analyzed by Liquid Chromatography tandem Mass Spectrometry. PUFAs will be classified based on their precursors and CYP450, COX, LOX pro-resolving pathways. In parallel, to identify the genes, polyA mRNAs extracted from transduced cells will be analyzed by RNA-Seq.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided